CLINICAL TRIAL: NCT01765894
Title: Influence of Moderate Exercise on Blood Glucose in Type 2 Diabetics and Healthy Controls.
Acronym: DIEGO
Status: Completed | Type: Observational
Sponsor: University of Copenhagen (Other)
Collaborators: Department of Biomedical Sciences (Ambiguous); XLab, Center of Healthy Aging (Unknown)
Responsible Party: Principal Investigator, Merethe Hansen, PhD student Merethe Hansen, University of Copenhagen
Other Study IDs: H-1-2012-074
Record Dates: First submitted 2012-11-30; First posted 2013-01-10 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2014-02

CONDITIONS: Type 2 Diabetes and Exercise
Keywords: glucose homeostasis; endogenous glucose production; moderate exercise; type 2 diabetes; metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity | interventions — Diet, Carbohydrate Loading

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood and plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Normal glucose tolerance subjects: Healthy controls. If any medication then paused 3 days prior to test days. BMI: 20-35. VO2max: 20-50. Age: 30-60 years All subjects perform same tests. - See protocol for description.
  Interventions: Other: 45 minutes of moderate exercise at the fasted state. Before test day 2: 3 days of carbohydrate loading.
- DM2: Type 2 diabetics in diet treatment or type 2 diabetics who have paused their oral medication for 3 whole days.
  Insulin treatment is an exclusion criteria. If any other medication then paused 3 days prior to test days.
  BMI: 20-35. VO2max: 20-50. Age: 30-60 years All subjects perform same tests. - See protocol for description.
  Interventions: Other: 45 minutes of moderate exercise at the fasted state. Before test day 2: 3 days of carbohydrate loading.
- DM2 + Metformin: Type 2 diabetics in metformin treatment. Insulin treatment is an exclusion criteria. If any other medication (besides from metformin) then paused 3 days prior to test days.
  BMI: 20-35. VO2max: 20-50. Age: 30-60 years All subjects perform same tests. - See protocol for description
  Interventions: Other: 45 minutes of moderate exercise at the fasted state. Before test day 2: 3 days of carbohydrate loading.

INTERVENTIONS:
Other: 45 minutes of moderate exercise at the fasted state. Before test day 2: 3 days of carbohydrate loading.
  Other Names: exercise performed at 60% of heart rate reserve.

SUMMARY:
Project description

Research project title:

Influence of moderate exercise on blood glucose in type 2 diabetics and healthy controls.

Project description and objective

Obesity is so widespread in Denmark that 47% of the population is classed as overweight (BMI>=25) and around 13% of the population is classed as obese (BMI>=30).

The strong correlation between obesity and type 2 diabetes (at least 2/3 of type 2 diabetics are overweight) has led to many studies which look at different forms of exercise for this group, because weight loss may improve the diabetes and even defer the onset of the disorder and in doing so lower complications and increase long term survival.

For people who do not have type 2 diabetes, the work-induced increased sympathetic activity will lead to suppressed insulin secretion and increased glucagon secretion. This increases the endogenous glucose production from the liver and thus maintains a normal concentration of blood sugar in a physical training situation where the demand for glucose has increased.

The theory behind the project is that the mechanisms that help to increase glucose production in the liver during physical activity are weaker in type 2 diabetics, which can cause hypoglycaemia during and after physical exercise. In other words, we want to study the liver's sensitivity to stimulus from physical work by patients with type 2 diabetes and in relevant healthy control subjects.

Previous studies have indicated that this type of mechanism is not intact in type 2 diabetics; because the level of insulin does not fall as expected during or after physical training. However, there are no existing studies that measure the liver's glucose secretion using stable isotopes during prolonged moderate physical work. Measuring this will help to clarify our understanding of glucose homeostasis in type 2 diabetics.

This study is very relevant, because it may be expected that the preferred form of physical exercise of an overweight type 2 diabetic can be of moderate intensity and previous studies also show that this form of physical exercise delivers health gains in terms of an improvement in insulin sensitivity and a reduction in the level of insulin.

The objective of this study is to determine if the level of blood glucose stays constant before, during and after physical training and to examine the liver's ability to secret glucose accordingly.

DETAILED DESCRIPTION:
Design

A group of 20 people with type 2 diabetes and 10 control subjects are twice invited to the laboratory, respectively.

The type 2 diabetes group consist of 10 individuals being treated with metformin and 10 individuals who are not being treated with Metformin. The latter group may be diet-treated diabetics or diabetics who have stopped taking their oral antidiabetic agent for 72 hours before the day of the experiment.

On the first visit, the following is carried out:

* DXA scan, blood pressure measurement, determination of ECG and VO2-max on a cycleergometer
* Blood sample
* Questionnaire about everyday physical activity (I-PAQ)

On the second visit, the following is carried out:

* 3 days of carbohydrate loading prior to this day.(By diet recommendations).
* Insertion of arterial cannula, blood sample extraction.
* Insertion of venus cannula. Insertion of stable glucose isotopes over a period of 4.5 hours: 2,5 hours of relaxation in bed followed by 45 minutes of cycling on an exercise bicycle (during continued isotope infusion) at 60% of maximum heart rate reserve, which was measured on test day 1. Followed by relaxation with continued blood sampling and isotope infusion, one hour after cycling ceased.

Inclusion criteria

* Age between 30 and 60 years old,
* Maximum oxygen consumption between 20 and 50 ml/kg/minute,
* BMI between 25 and 35 kg/m2,
* Normal ECG,
* Must have a stable weight throughout the last three months and have a normal balanced diet,
* Can cycle for 45 minutes

Exclusion criteria

* For patients with type 2 diabetes: insulin treatment,
* ECG that indicates cardiovascular disease,
* Illness or medicine that may affect the results,
* On-going weight loss diet

DXA scan

Minimal radiation - The scan lasts from six to 10 minutes and the total radiation dose with measuring is below 0.01 mSv (millisievert). This is approximately equivalent to the natural daily background exposure.

Cycling test

Prior to this test, an ECG is carried out and the person is quizzed about his/her state of health. Regarding all experiments, there is quick access to doctors in the laboratory. The laboratory is equipped with a defibrillator.

Infusion with stable glucose isotopes

Stable glucose isotopes occur naturally in the body, though in much smaller amounts. They are not radioactive and require no special precautions.

Blood sampling

An arterial cannula is inserted, from which blood samples are subsequently taken. A sample is immediately analysed (ABL analyser) for glucose and lactate concentrations and blood gases, Hgb and Hct.

Other blood samples are processed on a centrifuge and the plasma is frozen at - 80 °C until it will be analysed.

The plasma is analysed to determine concentrations of:

Insulin, glucagon, cortisol, growth hormone (GH), adrenocorticotrophic hormone (ACTH),C-peptide, catecholamines , alanin, concentration of ketone, cholesterol free fatty acids,glycerol, glucose isotope (Ra) content before, during and after the cycling.

The biological material (in the form of plasma) will be stored in a freezer. When the experiment is completed, the material will be analysed in our laboratories. When all of the analysis has been carried out, any excess materials will be destroyed. All materials will be stored anonymously.

Ethical considerations

At all times, the study will be carried out in accordance with the latest of Helsinki and current Danish legislation.

Among other things, this includes voluntary participation and that test subjects can withdraw their consent at any time and without having to provide any explanation.

The study protocol and the written patient information will be submitted to the Research Ethics Committee of the Capital Region of Denmark and the Danish Data Protection Agency will be informed. Patient inclusion cannot begin until a written approval has been received from both of these institutions. Both positive and, negative and inconclusive results must be published.

ELIGIBILITY:
Inclusion Criteria:

* Age between 30 and 60 years old
* Maximum oxygen consumption between 20 and 50 ml/kg/minute
* BMI between 25 and 35 kg/m2
* Normal ECG
* Must have a stable weight throughout the last three months and have a normal balanced diet
* Can cycle for 45 minutes

Exclusion Criteria:

* For patients with type 2 diabetes: insulin treatment
* ECG that indicates cardiovascular disease
* Illness or medicine that may affect the results
* On-going weight loss diet

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * 10 type 2 Diabetics without medication
  * 10 type 2 Diabetics on Metformin treatment
  * 10 matched healthy controls
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2012-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Glucose homeostasis in controls, type 2 diabetics without medication and type 2 diabetics in metformin treatment. | Observational study. Glucose homeostasis is tested one day only (in our Lab). Samples are taken 2,5 hours before, during and untill 1 hour after 45 minutes of exercise. Samples are taken every 5 minutes.
  Glucose, hormones, substrates, metabolites and glucose-isotopes as mentioned in the protocol.
  These end points will be measured on test day 2 only. Hormones and metabolites will be measured as AUC and total concentrations.

SECONDARY OUTCOMES:
MAP during moderate exercise | 45 min of moderate exercise (test day 2).
  MAP is continuously measured during exercise for 45 mins. (At 60% heart rate reserve)
vo2max | one measurement each subject (test day 1)
  Is measured in all subjects prior to test day 2
DXA-values | one measurement each subject (test day 1)
  DXA (fat%, lean body mass, BMD)is measured prior to test day 2
IL-6 and incretins | Observational study. Each test subject is tested for IL-6 and incretins one day only (in our Lab), where blood samples are taken continously during the test day every 5 minutes before, during and after exercise (test day 2).
  Effect of exercise on IL-6 and incretins. Described as AUC and total concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: Flemming Dela, professor, Principal Investigator — University of Copenhagen
Locations (1):
- XLab, Center for Healthy Aging, Department of Biomedical Sciences, University of Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Derived] Hansen M, Palsoe MK, Helge JW, Dela F. The effect of metformin on glucose homeostasis during moderate exercise. Diabetes Care. 2015 Feb;38(2):293-301. doi: 10.2337/dc14-1480. Epub 2014 Dec 2. PMID 25468944